CLINICAL TRIAL: NCT07266688
Title: Evaluation of the Efficacy and Safety of Treatment With a Medical Device Containing Pistacia Lentiscus in Patients With Vasomotor Rhinitis: A Multicenter, Prospective, Randomized, Controlled Clinical Trial
Brief Title: Evaluation of Bactorinol® Nasal Spray in Adult Patients With Vasomotor Rhinitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: University of Urbino "Carlo Bo" (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116/22.11.2024/BACTORINOL
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Vasomotor Rhinitis
MeSH Terms: conditions — Rhinitis, Vasomotor

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group, randomized controlled design with 1:1 allocation to Bactorinol® nasal spray or isotonic saline solution.
Masking Description: Open-label study; no masking of participants or investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bactorinol® Nasal Spray (Treatment Arm) (Experimental): Participants receive Bactorinol® nasal spray containing winterized Pistacia lentiscus oil (medical device). Dosage: 3 puffs per nostril, three times daily for 20 consecutive days.
  Interventions: Device: Bactorinol® Nasal Spray
- Isotonic Saline Solution (Control Arm) (Active Comparator): Participants receive isotonic saline solution nasal spray. Dosage: 3 administrations per nostril, three times daily for 20 consecutive days.
  Interventions: Other: Isotonic Saline Solution

INTERVENTIONS:
Device: Bactorinol® Nasal Spray — Bactorinol® nasal spray containing winterized Pistacia lentiscus oil. Administered as 3 puffs per nostril, three times daily for 20 consecutive days.
  Other Names: Winterized Pistacia lentiscus oil nasal spray
  Arms: Bactorinol® Nasal Spray (Treatment Arm)
Other: Isotonic Saline Solution — Isotonic saline nasal spray administered as 3 sprays per nostril, three times daily for 20 consecutive days.
  Other Names: Normal saline nasal spray (Control)
  Arms: Isotonic Saline Solution (Control Arm)

SUMMARY:
This study aims to evaluate the effectiveness and safety of Bactorinol® nasal spray, a medical device containing winterized Pistacia lentiscus oil, in adults with vasomotor rhinitis. Vasomotor rhinitis is a chronic condition characterized by nasal congestion, rhinorrhea, and impaired nasal airflow.

In this multicenter, prospective, randomized, controlled clinical trial, 100 adult participants will be assigned in a 1:1 ratio to receive either Bactorinol® nasal spray or isotonic saline solution for 20 consecutive days. The primary objective is to determine whether Bactorinol® improves nasal airflow, measured by Peak Nasal Inspiratory Flow (PNIF). Secondary objectives include evaluating changes in symptoms and quality of life using the SNOT-22 questionnaire, assessing nasal cytology, and monitoring treatment compliance and adverse events.

The results of this study may help identify a non-pharmacological, natural-extract-based treatment option for patients with vasomotor rhinitis.

DETAILED DESCRIPTION:
Vasomotor rhinitis is a chronic inflammatory condition of the nasal mucosa characterized by airflow obstruction, dysregulated mucus production, and impaired mucociliary clearance. Environmental factors, mucosal dryness, and alterations in epithelial function contribute to symptoms, and current treatment options are often limited or unsatisfactory.

Bactorinol® nasal spray is a medical device formulated with winterized Pistacia lentiscus oil, which contains terpenes and polyphenols with recognized emollient, anti-inflammatory, antibacterial, and antibiofilm properties. These characteristics may help reduce mucosal irritation, improve mucociliary function, and relieve nasal congestion.

This multicenter, prospective, randomized, controlled, parallel-group clinical trial will enroll 100 adults with a confirmed diagnosis of vasomotor rhinitis. Participants will be randomized 1:1 to receive either Bactorinol® nasal spray (3 puffs per nostril, three times daily) or isotonic saline solution with the same dosing schedule, for 20 days.

The primary endpoint is the change in nasal airflow as measured by Peak Nasal Inspiratory Flow (PNIF) from baseline to the end of treatment. Secondary assessments include changes in quality of life measured by the SNOT-22 questionnaire, nasal cytology via rhinocytogram, treatment compliance, and adverse events. Clinical and cytological evaluations will be performed at baseline and at the end of the 20-day treatment period.

The study is designed to determine whether Bactorinol® provides clinically meaningful improvement in nasal breathing and symptom burden in patients with vasomotor rhinitis and to assess its safety and tolerability when used as directed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 to 70 years.
* Confirmed diagnosis of vasomotor rhinitis.
* Ability to understand the study procedures and provide written informed consent.
* Ability to follow study instructions.
* Availability to undergo scheduled evaluations.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Stenosing deviation of the nasal septum.
* Current or recurrent episodes of epistaxis.
* History of nasal endoscopic surgery within the past 6 months.
* Use of systemic antibiotics within the previous 30 days.
* Known hypersensitivity to any component of the study products.
* Concomitant topical medications applied to the nasal mucosa.
* Participation in another clinical trial or completion of another trial within the last month.
* Failure or unwillingness to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Change in Peak Nasal Inspiratory Flow (PNIF) | 20 days
  PNIF will be measured using a Peak Nasal Inspiratory Flow meter to assess nasal airflow. The value at baseline (Visit 1) will be compared with the value at the end of treatment (Visit 2).

SECONDARY OUTCOMES:
Change in Quality of Life Measured by SNOT-22 | 20 days
  Quality of life will be assessed using the validated Sino-Nasal Outcome Test (SNOT-22) questionnaire at baseline and at the end of treatment.
Change in Nasal Cytology (Rhinocytogram) | 20 days
  Nasal cytology will be evaluated using a rhinocytogram, assessing quantitative and semi-quantitative cellular components including neutrophils, metachromatic cells, goblet cells, eosinophils, mast cells, bacteria, spores/fungi, and presence of biofilm.
Treatment Compliance | 20 days
  Compliance will be assessed by counting returned product at the end of treatment and verifying the number of nebulizations performed.
Incidence of Adverse Events | 20 days
  All adverse events reported by participants or observed by investigators during the study period will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Urbino Carlo Bo, Urbino, Pesaro E Urbino, Italy

IPD SHARING:
Plan to Share IPD: No